CLINICAL TRIAL: NCT05838495
Title: A Single-center, Open-label Study on the Nutritional Adequacy, Tolerability, and Safety of a Hypercaloric, Plant-based, Real Food Ingredient Formula for Tube Fed Pediatric Patients
Brief Title: Nutritional Tolerance and Safety of a Tube Feeding Formula in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: N02-20-01-T0004; 22.01.CA.HCN (Other: Sponsor)
Record Dates: First submitted 2023-04-05; First posted 2023-05-01 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Enteral Feeding

STUDY DESIGN:
Intervention Model Description: Prospective, single arm, non-randomized, open-label, observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enteral tube fed children (Experimental): Children being fed an enteral formula with a feeding tube
  Interventions: Other: formulated liquid diet

INTERVENTIONS:
Other: formulated liquid diet — will be fed exclusively the pediatric enteral study formula with a feeding tube

SUMMARY:
To assess the efficacy, tolerance, and safety of a pediatric enteral formula in children.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy (ability to meet prescribed calorie and protein needs), tolerance, and safety of a pediatric enteral formula (i.e., the study product) in participants aged 1-13 years for 14 days of use.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable, enterally tube-fed children
* Aged 1 to 13 years (inclusive) at the time of screening.
* Currently tolerating enteral feeding and should be appropriate for study formula
* Requires enteral tube feeding to provide 90% or more of their nutritional needs
* signed informed consent

Exclusion Criteria:

* Has a condition which contraindicates enteral feeding (e.g., intestinal obstruction).
* Currently using or has previously used the study product
* Any medical condition or contraindicated medications that would contraindicate use of the study product
* Any illness within ~5-7 days of screening and/or baseline lasting >48 hours and assessed by the PI to have affected nutritional intake on a case-by-case basis.
* Participation in another interventional clinical study
* Any condition or abnormality that, in the opinion of the PI, would compromise the safety of the participant or the quality of the study data.

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-06 (Actual)

PRIMARY OUTCOMES:
Nutritional efficacy - energy | 14 days
  Percent of daily calorie nutritional goals met

SECONDARY OUTCOMES:
Nutritional efficacy - protein | 14 days
  Percent of daily protein nutritional goals met
Frequency of nausea | 14 days
  Daily frequency of nausea for each participant
Frequency of vomiting | 14 days
  Daily frequency of vomiting for each participant
Bristol Stool Chart | 14 days
  Daily reporting of stool parameters using Bristol stool chart. Scale from 1-7. Type 1: Separate hard lumps (hard to pass) Type 2: Lumpy, hard, sausage-shaped Type 3: Sausage-shaped with cracks on the surface Type 4: Sausage-shaped or snake-like; smooth and soft Type 5: Soft blobs with clear-cut edges (easy to pass) Type 6: Fluffy pieces with ragged edges; mushy Type 7: Entirely liquid, watery, no solid pieces
Adverse events | 14 days
  Daily adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Hulst, MD, Principal Investigator — The Hospital for Sick Children; Cindy Steel, MSc, Study Chair — Nestle Health Science Canada; Krys Araujo Torres, MD, Study Director — Nestle Health Science USA
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No